CLINICAL TRIAL: NCT00030732
Title: Gemcitabine Plus Capecitabine Versus Gemcitabine Alone In Advanced Pancreatic Cancer. A Randomized Phase III Trial
Brief Title: Gemcitabine With or Without Capecitabine in Treating Patients With Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Collaborators: Central European Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 44/00; SWS-SAKK-44/00 (Other: SAKK); CECOG/PAN-1.3.001; EU-20142
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Pancreatic Cancer
Keywords: stage III pancreatic cancer; recurrent pancreatic cancer; adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemcitabine + Capecitabine (Active Comparator): Gemcitabine + Capecitabine
  Interventions: Drug: Gemcitabine + Capecitabine
- Gemcitabine alone (Active Comparator): Gemcitabine alone
  Interventions: Drug: Gemcitabine alone

INTERVENTIONS:
Drug: Gemcitabine + Capecitabine — Gemcitabine + Capecitabine
  Arms: Gemcitabine + Capecitabine
Drug: Gemcitabine alone — Gemcitabine alone
  Arms: Gemcitabine alone

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known if gemcitabine is more effective with or without capecitabine in treating pancreatic cancer.

PURPOSE: Randomized phase III trial to determine the effectiveness of gemcitabine with or without capecitabine in treating patients who have advanced pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival of patients with advanced pancreatic cancer treated with gemcitabine with or without capecitabine.
* Compare the clinical benefit response, objective tumor response, duration of response, and time to progression in patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to metastases (yes vs no), pain (yes vs no), Karnofsky performance status (60-80% vs 90-100%), and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive gemcitabine IV over 30 minutes on days 1 and 8 and oral capecitabine twice daily on days 1-14. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients initially receive gemcitabine IV over 30 minutes weekly for 7 weeks. After 1 week of rest, patients receive gemcitabine IV over 30 minutes weekly for 3 weeks. Treatment then repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, weekly for weeks 2-7, and then before each gemcitabine administration.

Patients are followed every 9 weeks.

PROJECTED ACCRUAL: A total of 300 patients (150 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed primary inoperable or metastatic pancreatic adenocarcinoma
* No CNS metastases

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10.0 g/dL

Hepatic:

* Bilirubin no greater than 5 times normal
* AST/ALT no greater than 5 times normal
* Alkaline phosphatase no greater than 5 times normal

Renal:

* Creatinine clearance at least 30 mL/min

Gastrointestinal:

* No grade 2 or greater nausea or grade 1 or greater vomiting
* No medical condition that would interfere with taking oral medications or with gastrointestinal absorption (e.g., small bowel obstruction)

Other:

* No prior unanticipated severe reaction to fluoropyrimidine therapy
* No known hypersensitivity to fluorouracil
* No known dihydropyrimidine dehydrogenase deficiency
* No active infection
* No other serious concurrent systemic disorders that would preclude study participation
* No other malignancy within the past 5 years except adequately treated carcinoma in situ of the cervix or basal cell skin cancer
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior capecitabine
* No prior chemotherapy for advanced pancreatic cancer
* At least 1 year since prior radiochemotherapy for pancreatic cancer

Endocrine therapy:

* Not specified

Radiotherapy:

* See Chemotherapy
* At least 1 year since prior adjuvant radiotherapy for pancreatic cancer
* No concurrent radiotherapy

Surgery:

* Prior Whipple procedure or duodenal bypass allowed

Other:

* At least 1 month since prior investigational agents
* No concurrent sorivudine or its chemically related analogues (e.g., brivudine)
* No other concurrent anticancer or investigational drugs

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2001-06; Primary Completion 2004-06 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Gemcitabine + Capecitabine vs. Gemcitabine alone | 8 weeks
  To compare survival, efficacy, quality of life and toxicity between the combination therapy (Capecitabine and Gemcitabine) and the monotherapy (Gemcitabine alone) in advanced pancreatic cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Herrmann, MD, Study Chair — Universitaetsspital-Basel; Werner Scheithauer, MD, Study Chair — Allgemeines Krankenhaus - Universitatskliniken
Locations (18):
- Allgemeines Krankenhaus der Stadt Wien, Vienna, Austria
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel
- Italy (2):
  - Istituto Nazionale per lo Studio e la Cura dei Tumori, Milan
  - Istituto Nazionale per lo Studio e la Cura dei Tumori, Naples
- Switzerland (14):
  - Kantonspital Aarau, Aarau
  - Saint Claraspital AG, Basel
  - Universitatsspital-Basel, Basel
  - Inselspital, Bern, Bern
  - Spitalzentrum Biel, Biel
  - Ratisches Kantons und Regionalspital, Chur
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Institut Central des Hopitaux Valaisans, Sion
  - Regionalspital, Thun
  - City Hospital Triemli, Zurich
  - Oncology Institute of Southern Switzerland, Zurich
  - UniversitaetsSpital, Zurich

REFERENCES:
- [Result] Bernhard J, Dietrich D, Glimelius B, Hess V, Bodoky G, Scheithauer W, Herrmann R. Estimating prognosis and palliation based on tumour marker CA 19-9 and quality of life indicators in patients with advanced pancreatic cancer receiving chemotherapy. Br J Cancer. 2010 Oct 26;103(9):1318-24. doi: 10.1038/sj.bjc.6605929. Epub 2010 Sep 28. PMID 20877359
- [Result] Bernhard J, Dietrich D, Scheithauer W, Gerber D, Bodoky G, Ruhstaller T, Glimelius B, Bajetta E, Schuller J, Saletti P, Bauer J, Figer A, Pestalozzi BC, Kohne CH, Mingrone W, Stemmer SM, Tamas K, Kornek GV, Koeberle D, Herrmann R; Central European Cooperative Oncology Group. Clinical benefit and quality of life in patients with advanced pancreatic cancer receiving gemcitabine plus capecitabine versus gemcitabine alone: a randomized multicenter phase III clinical trial--SAKK 44/00-CECOG/PAN.1.3.001. J Clin Oncol. 2008 Aug 1;26(22):3695-701. doi: 10.1200/JCO.2007.15.6240. PMID 18669454
- [Result] Hess V, Glimelius B, Grawe P, Dietrich D, Bodoky G, Ruhstaller T, Bajetta E, Saletti P, Figer A, Scheithauer W, Herrmann R. CA 19-9 tumour-marker response to chemotherapy in patients with advanced pancreatic cancer enrolled in a randomised controlled trial. Lancet Oncol. 2008 Feb;9(2):132-8. doi: 10.1016/S1470-2045(08)70001-9. PMID 18249033
- [Result] Herrmann R, Bodoky G, Ruhstaller T, Glimelius B, Bajetta E, Schuller J, Saletti P, Bauer J, Figer A, Pestalozzi B, Kohne CH, Mingrone W, Stemmer SM, Tamas K, Kornek GV, Koeberle D, Cina S, Bernhard J, Dietrich D, Scheithauer W; Swiss Group for Clinical Cancer Research; Central European Cooperative Oncology Group. Gemcitabine plus capecitabine compared with gemcitabine alone in advanced pancreatic cancer: a randomized, multicenter, phase III trial of the Swiss Group for Clinical Cancer Research and the Central European Cooperative Oncology Group. J Clin Oncol. 2007 Jun 1;25(16):2212-7. doi: 10.1200/JCO.2006.09.0886. PMID 17538165
- [Result] Gargiulo P, Dietrich D, Herrmann R, Bodoky G, Ruhstaller T, Scheithauer W, Glimelius B, Berardi S, Pignata S, Brauchli P. Predicting mortality and adverse events in patients with advanced pancreatic cancer treated with palliative gemcitabine-based chemotherapy in a multicentre phase III randomized clinical trial: the APC-SAKK risk scores. Ther Adv Med Oncol. 2019 Jan 2;11:1758835918818351. doi: 10.1177/1758835918818351. eCollection 2019. PMID 30636977